CLINICAL TRIAL: NCT06265428
Title: A Phase III, Multicenter, Open-label, Randomized Study to Compare DB-1303 Versus T-DM1 in Patients With HER2-positive Unresectable/Metastatic Breast Cancer Who Have Been Treated With Trastuzumab and a Taxane (Dynasty-Breast01)
Brief Title: A Study to Compare DB-1303/BNT323 Versus T-DM1 in Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB-1303-O-3001; CTR20233403 (Other: CENTER FOR DRUG EVALUATION, NMPA)
Record Dates: First submitted 2024-01-05; First posted 2024-02-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive; Breast Cancer; BC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DB-1303/BNT323 (Experimental): Enrolled patients will receive DB-1303/BNT323 by intravenous (I.V.) infusion
  Interventions: Drug: DB-1303/BNT323
- T-DM1 (Experimental): Enrolled patients will receive T-DM1 by I.V. infusion
  Interventions: Drug: T-DM1

INTERVENTIONS:
Drug: DB-1303/BNT323 — Administered I.V.
  Arms: DB-1303/BNT323
Drug: T-DM1 — Administered I.V.
  Arms: T-DM1

SUMMARY:
This study is designed to compare efficacy and safety of DB-1303/BNT323 versus T-DM1 in HER2-positive, unresectable and/or metastatic breast cancer patients previously treated with trastuzumab and taxane.

DETAILED DESCRIPTION:
This is a randomized controlled, 2-arm, open-label, multicenter phase III study to assess the efficacy and safety of DB-1303/BNT323 versus Trastuzumab Emtansine (T-DM1) in patients with human epidermal growth factor receptor 2 (HER2) -positive unresectable/metastatic breast cancer who have been treated with trastuzumab and taxanes. Approximately 224 patients with unresectable or metastatic HER2-positive breast cancer will be randomized 1:1 to receive DB-1303/BNT323 or T-DM1, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ≥ 18 years at the time of voluntary signing of informed consent.
* Pathologically confirmed unresectable or metastatic HER2 positive breast cancer previously treated with trastuzumab and taxane
* Eastern Cooperative Oncology Group (ECOG) performance status score is 0 or 1.
* Presence of at least one measurable lesion according to RECIST v1.1
* Expected survival time ≥ 12 weeks.
* Patients must give informed consent to this study and voluntarily sign written informed consent form prior to the study.

Exclusion Criteria:

* Prior anti-HER2 ADC therapy.
* Previous history of interstitial lung disease/noninfectious pneumonitis/radiation pneumonitis requiring steroid therapy.
* Known serious hypersensitivity to the active ingredients of the study drug, inactive ingredients in the formulation, or other antibody drugs.
* Multiple primary malignancies within 3 years, except for adequately resected non-melanoma skin cancer, curatively treated in situ tumor, or contralateral breast cancer
* Uncontrolled infection requiring intravenous antibiotics, antiviral or antifungal agents, autoimmune disease requiring treatment, uncontrolled diabetes, hypertension, or other systemic disease that makes compliance with study procedures difficult
* Unrecovered toxicity from prior anticancer therapy, defined as toxicity (except for alopecia) not recovered to ≤Grade 1 (NCI-CTCAE v5.0) or baseline.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by Blinded Independent Central Review (BICR) assessment per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 24 months.
  Defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by BICR or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 24 months.
  Defined as the time from randomization to death due to any cause.
Progression Free Survival (PFS) by Investigator assessment per RECIST 1.1 | Up to approximately 24 months.
  Defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by investigator or death due to any cause, whichever occurs first.
Objective response rate (ORR) by BICR and investigator assessment per RECIST 1.1 | Up to approximately 24 months.
  Defined as the percentage of patients who have a complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by BICR and investigator assessment.
Duration of response (DoR) by BICR and investigator assessment per RECIST 1.1 | Up to approximately 24 months.
  Defined as the time from first response (CR or PR) to subsequent disease progression per RECIST 1.1 as assessed by BICR and investigator assessment, or death from any cause, whichever occurs first.
PK parameters: maximum observed concentration (Cmax) | Up to approximately 24 months.
  Maximum observed concentration (Cmax) of DB-1303/BNT323 Antibody-drug conjugate (ADC) and free toxin P1003, etc. after DB-1303/BNT323 administration
PK parameters: time to maximum concentration (Tmax) | Up to approximately 24 months.
  Time to maximum concentration (Tmax) of DB-1303/BNT323 ADC and free toxin P1003, etc. after DB-1303/BNT323 administration
Adverse events (AEs) | Up to approximately 24 months.
  Number and percentage of patients who report serious adverse events (SAEs), treatment-emergent adverse events (TEAEs), TEAEs leading to study drug discontinuation, adverse events of special interest (AESIs) (graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0[NCI-CTCAE v5.0])
Patient reported outcomes (PROs): European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) - C30 | Up to approximately 24 months.
  Change from baseline in the functioning/symptom/global quality of life (QoL) subscales of EORTC QLQ-C30. Scale scores range from 0-100. For functioning and global QoL scales, higher scores indicate better functioning or global health status. For symptom scales, higher scores indicate greater symptom burden.
Patient reported outcomes (PROs): EORTC QLQ-BR45 | Up to approximately 24 months.
  Change from baseline in the functioning/symptom subscales of EORTC QLQ-BR45. Scale scores range from 0-100. For functioning scales, higher scores indicate better functioning. For symptom scales, higher scores indicate greater symptom burden.
Patient reported outcomes (PROs): European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) | Up to approximately 24 months.
  Change from baseline in EQ-5D-5L health state utility index score and Visual Analogue Scale (VAS) score. VAS score range from 0-100, higher scores indicate better health status.
European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) | Up to approximately 24 months.
  EQ-5D-5L health state utility index score and Visual Analogue Scale (VAS) score. The change from baseline value will be reported.
Anti-drug antibodies (ADA) | Up to approximately 24 months.
  Number and percentage of patients who develop anti-drug antibody (ADA) for DB-1303/BNT323.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hu, Study Director — DualityBio Inc.
Locations (48):
- China (48):
  - 015, Bengbu, Anhui
  - 016, Hefei, Anhui
  - 029, Hefei, Anhui
  - 001, Beijing, Beijing Municipality
  - 010, Beijing, Beijing Municipality
  - 038, Jilin, Changchun
  - 036, Fuzhou, Fujian
  - 037, Xiamen, Fujian
  - 023, Guangzhou, Guangdong
  - 024, Guangzhou, Guangdong
  - 026, Guangzhou, Guangdong
  - 028, Huizhou, Guangdong
  - 017, Nanning, Guangxi
  - 022, Nanning, Guangxi
  - 043, Haikou, Hainan
  - 045, Baoding, Hebei
  - 048, Shijiazhuang, Hebei
  - 020, Haerbin, Heilongjiang
  - 018, Luoyang, Henan
  - 006, Zhengzhou, Henan
  - 005, Zhengzhou, Henan
  - 011, Wuhan, Hubei
  - 009, Wuhan, Hubei
  - 030, Changsha, Hunan
  - 027, Nanjing, Jiangsu
  - 004, Nanjing, Jiangsu
  - 044, Xuzhou, Jiangsu
  - 014, Nanchang, Jiangxi
  - 008, Changchun, Jilin
  - 032, Dalian, Liaoning
  - 040, Binzhou, Shandong
  - 031, Jinan, Shandong
  - 047, Jinan, Shandong
  - 012, Linyi, Shandong
  - 039, Yantai, Shandong
  - 002, Shanghai, Shanghai Municipality
  - 046, Shanghai, Shanghai Municipality
  - 035, Taiyuan, Shanxi
  - 003, Xi’an, Shanxi
  - 007, Chengdu, Sichuan
  - 041, Neijiang, Sichuan
  - 034, Yibin, Sichuan
  - 021, Tianjin, Tianjin Municipality
  - 013, Ürümqi, Xinjiang
  - 033, Kunming, Yunnan
  - 019, Hangzhou, Zhejaing
  - 025, Hangzhou, Zhejiang
  - 042, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No